CLINICAL TRIAL: NCT03156114
Title: An Open Label, Phase I Dose-finding Study of BI 754111 in Combination With BI 754091 in Patients With Advanced Solid Cancers Followed by Expansion Cohorts at the Selected Dose of the Combination in Patients With Non-small Cell Lung Cancer and Other Solid Tumors
Brief Title: This Study Tests the New Medicine BI 754111 Alone or in Combination With Another New Substance BI 754091 in Patients With Advanced Cancer. The Study Tests Different Doses to Find the Best Dose for Continuous Treatment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1381-0002; 2017-005042-29 (EudraCT Number)
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose escalation cohort: BI 754111 4 mg + 240 mg ezabenlimab (Experimental): 4 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 20 mg + 240 mg ezabenlimab (Experimental): 20 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 80 mg + 240 mg ezabenlimab (Experimental): 80 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 200 mg + 240 mg ezabenlimab (Experimental): 200 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 400 mg + 240 mg ezabenlimab (Experimental): 400 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 600 mg + 240 mg ezabenlimab (Experimental): 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose escalation cohort: BI 754111 800 mg + 240 mg ezabenlimab (Experimental): 800 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose-Expansion Cohort G (Experimental): 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w) in patients with 2nd and 3rd line Non-small cell lung cancer (NSCLC) who progressed on anti-programmed cell death 1 (PD-1) or anti-programmed cell death ligand 1 (PD-L1) treatment.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose-Expansion Cohort H (Experimental): 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w) in ≥2nd line microsatellite stable anti-PD-1 and anti-PD-L1 treatment-naïve metastatic colorectal cancer (mCRC).
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose-Expansion Cohort I (Experimental): 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w) in patients with any solid tumour with high tumour mutational burden (TMB) and/or microsatellite instability high (MSI-H) and/or DNA mismatch repair deficient solid tumours who have received 1 prior anti-PD-1 or anti-PD-L1 treatment regimen.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Dose-Expansion Cohort J (Experimental): 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w) patients with 1st line epidermal growth factor receptor (EGFR) wildtype (WT) and anaplastic lymphoma kinase (ALK) wildtype NSCLC. Patients may have any level of PD-L1 expression, but only a maximum of 10 patients with PD-L1 high expression (≥50% PD-L1) were enrolled.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111

INTERVENTIONS:
Drug: Ezabenlimab — 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w)
Drug: BI 754111 — Different dosages of BI 754111 given as an intravenous infusion on day 1 of 21-day cycles (q3w).

SUMMARY:
This is a study in adults with advanced solid tumors including non-small cell lung cancer.

The study tests the combination of two medicines called BI 754111 and BI 754091 that may help the immune system to fight the cancer. Such medicines are called immune checkpoint inhibitors.

The study has two parts. In the first part, doctors want to find out the highest dose of 2 medicines that people with solid tumors can tolerate. This dose is then used for the second part of the study.

In the second part, the combination of the two medicines is tested in patients with non-small cell lung cancer and other types of solid cancer. These patients had gotten treatment with anti-PD-1 or anti-PD-L1 medicines but their tumors have come back. The doctors check whether the combination of BI 754111 and BI 754091 makes tumors shrink.

Both medicines are given as an infusion into the vein every 3 weeks. If there is benefit for the patients and if they can tolerate it, the treatment is given for maximum of 1 year. During the entire study doctors will regularly check the health of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written Informed consent form (ICF) prior to any trial-specific procedures, sampling, or analyses
* Patients ≥18 years of age at the time of signature of the ICF
* Part I (dose escalation):

  --Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours (any type)
  * For whom no therapy of proven efficacy exists, or who are not amenable to standard therapies.
  * Must have measurable lesions according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
  * Previous treatment with an anti-programmed cell death 1 (receptor) (PD-1) monoclonal antibody (mAb) is allowed as long as the last administration of the anti-PD-1 mAb on the previous treatment is a minimum of 60 days prior to starting treatment in this trial.
* Part II (dose expansion):

  * Patients must have measurable disease per RECIST v1.1 criteria, must have at least 1 tumour lesion amenable to biopsy, and must be medically fit and willing to undergo a biopsy before first treatment (if adequate archival tissue is not available) and, unless clinically contraindicated, after 6 weeks on therapy.
  * Dose Expansion Cohorts: Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours of one of the following types:

    * Second and 3rd line Non-small cell lung cancer (NSCLC) patients:

      * Must have progressed on anti-PD-1 or anti-programmed cell death ligand 1 (PD-L1) treatment after having achieved radiologically confirmed benefit (minimum of stable disease)
      * Must have had a minimum duration of benefit of 4 months and minimum treatment duration of 2 months on the previous anti- PD-1 or anti-PD-L1 treatment without experiencing disease progression during that period.
      * The anti-PD-1- or anti-PD-L1-containing treatment must have been the latest treatment regimen prior to enrolling in this trial
      * Must be within >4 and <12 weeks since the latest treatment and their first dose in this trial. Patients who have had anti-PD-1 or anti-PD-L1 monotherapy as their first-line NSCLC treatment regimen must have a PD-L1 expression level of ≥1% at baseline (local validated testing).
    * Anti-PD-1 or anti-PD-L1 treatment-naïve patients with microsatellite stable Metastatic colorectal Cancer (mCRC):

      * Patients must have had ≥ 1 line treatment
      * Must have microsatellite stable disease (identified using any validated test)
      * Must be anti-PD-1 and anti-PD-L1 treatment naïve
    * Anti-PD-1 or anti-PD-L1 pretreated patients with any high Tumour mutational burden (TMB) (≥10 mutations/Mb) and/or Microsatellite instability high (MSI-H) and/or DNA MMRd solid tumours

      * Patients must have high TMB (≥ 10 mutations/Mb) and/or MSI-H and/or DNA mismatch repair deficient (MMRd) (measured using any validated test).
      * Patients must have received 1 prior anti-PD-1 or anti-PD-L1 treatment regimen.
    * 1st-line squamous or non-squamous NSCLC patients:

      * Patients must be treatment naïve
      * Must be epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) wild type (only applicable to patients with non-squamous NSCLC)
      * Regardless of PD-L1 expression level. However, the number of patients with high level of PD-L1 expression (≥50% PD-L1) will be limited to a maximum of 10 patients
* Eastern Cooperative Oncology Group (ECOG, R01-0787) score: 0 to 1
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control (that result in a low failure rate of less than 1% per year when used consistently and correctly) during trial participation and for at least 6 months after the last administration of trial medication. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Major surgery (major according to the Investigator's assessment) performed within 12 weeks prior to first trial treatment or planned within 12 months after screening, e.g., hip replacement
* Patients who must or wish to continue the intake of restricted medications (see Section 4.2.2.2) or any drug considered likely to interfere with the safe conduct of the trial
* Previous enrolment in this trial
* Any investigational or anti-tumour treatment, except BI 754091, within 4 weeks or within 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment.
* Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 neuropathy due to prior platinum-based therapy
* Prior treatment with anti-Lymphocyte-activation gene 3 (LAG-3) agents
* Patients with NSCLC that has EGFR mutations or ALK rearrangements (only applicable to patients with non-squamous NSCLC).
* Presence of other active invasive cancers other than the one treated in this trial within 5 years prior to screening, with the exception of appropriately treated basal-cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or other local tumours considered cured by local treatment
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of PD by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases.
* Inadequate organ function or bone marrow reserve as demonstrated by the laboratory values presented in Table 3.3.3: 1.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
  * Patients with an ejection fraction (EF) <55% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram, multi-gated acquisition scan). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
* History of pneumonitis within the last 5 years
* History of severe hypersensitivity reactions to other mAbs
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment.
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy
* Active infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at start of treatment in this trial
* Known history of human immunodeficiency virus infection or an active hepatitis B or C virus infection
* Interstitial lung disease
* Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes him/her an unreliable trial subject, unlikely to complete the trial, or unable to comply with the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - University of Miami, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Poland (2):
  - BioVirtus Research Site Sp. z o.o., Józefów
  - Oncology Center-Maria Sklodowska-Curie Institute, Warsaw
- Spain (4):
  - Hospital Universitari Dexeus, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Politècnic La Fe, Valencia
- Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Zettl M, Wurm M, Schaaf O, Mostbock S, Tirapu I, Apfler I, Lorenz IC, Frego L, Kenny C, Thibodeau M, Oquendo Cifuentes E, Reschke M, Moll J, Kraut N, Vogt A, Sedgwick JD, Waizenegger IC. Combination of two novel blocking antibodies, anti-PD-1 antibody ezabenlimab (BI 754091) and anti-LAG-3 antibody BI 754111, leads to increased immune cell responses. Oncoimmunology. 2022 Jun 16;11(1):2080328. doi: 10.1080/2162402X.2022.2080328. eCollection 2022. PMID 35756842
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an an open label, Phase I dose-finding study in patients with advanced solid cancers followed by expansion cohorts at the selected dose of the combination in patients with non-small cell lung cancer and other solid tumors.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Started | 4 | 9 | 9 | 9 | 9 | 9 | 6 | 21 | 40 | 39 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 9 | 9 | 9 | 9 | 6 | 21 | 40 | 39 | 17
Not completed — Other than listed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Subject decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Non-compliant with study drug | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 3 | 7 | 5 | 4
Not completed — Progressive disease | 4 | 8 | 8 | 5 | 8 | 6 | 5 | 17 | 31 | 27 | 7
Not completed — Currently on treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Treated Set (TS) included all patients who received at least 1 dose of BI 754111 or ezabenlimab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J | Total
Number analyzed (Participants) | 4 | 9 | 9 | 9 | 9 | 9 | 6 | 21 | 40 | 39 | 17 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.7) | 62.3 (10.8) | 61.8 (5.5) | 59.6 (19.2) | 59.9 (9.6) | 54.2 (6.2) | 60.2 (14.2) | 66.1 (7.9) | 55.4 (13.0) | 64.6 (11.1) | 71.5 (9.0) | 61.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 5 | 6 | 3 | 5 | 2 | 8 | 13 | 22 | 8 | 81
  Male | 3 | 1 | 4 | 3 | 6 | 4 | 4 | 13 | 27 | 17 | 9 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 7
  Not Hispanic or Latino | 4 | 9 | 8 | 9 | 7 | 8 | 4 | 20 | 38 | 36 | 15 | 158
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 6
  White | 4 | 9 | 8 | 6 | 6 | 8 | 4 | 20 | 36 | 34 | 16 | 151
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Maximum-tolerated Dose (MTD) of the BI 754111 Plus Ezabenlimab Combination
Description: The MTD is defined as the highest dose with less than 25% risk of the true Dose-limiting toxicity (DLT) rate being above 33%. DLTs include:
  Haematologic toxicities:
  * Any Grade 5 toxicity
  * Neutropenia ≥ Grade 4 for >5 days
  * Any duration febrile neutropenia
  * Grade 4 thrombocytopenia or Grade 3 with bleeding/platelet transfusion need
  * Unexplained Grade 4 anaemia.
  Non-haematological toxicities:
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3x Upper limit of normal (ULN) and total bilirubin >2x ULN without cholestasis signs
  * ≥Grade 4 AST or ALT of any duration
  * Any ≥Grade 3 non-haematologic toxicity with exceptions
  * Any Grade 4 or 5 adverse event (AE)
  * Any Grade 2 pneumonitis
  * Any Grade 2 uveitis, eye pain, or blurred vision not improving to Grade 1 within 2 weeks or requiring systemic treatment
  * Any ≥ Grade 2 toxicity causing inability to administer BI 754091 on Cycle 2 Day 1.
Time Frame: First treatment cycle, the first 21 days following the start of trial medication.
Population: The MTD evaluation set included all patients in the dose escalation cohort who received BI 754111 or ezabenlimab, and who were not replaced within the MTD evaluation period (First treatment cycle, the first 21 days following the start of trial medication).
Measure: Number; unit: Milligram
Groups:
- Dose Escalation Cohort: BI 754111 + Ezabenlimab: Comprises all dose cohorts during the dose escalation phase. BI 754111 and ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w).
Arm/Group | Dose Escalation Cohort: BI 754111 + Ezabenlimab
Number analyzed (Participants) | 55
Milligram | NA — There were no dose-limiting toxicities experienced by any dose escalation cohort patient during the MTD evaluation period, thus MTD was not reached.

2. Primary Outcome: Dose Escalation: Number of Patients Experiencing DLTs During the Combination MTD Evaluation Period
Description: Number of patients experiencing DLTs during the combination MTD evaluation period (first cycle of BI 754111 plus ezabenlimab combination therapy) in patients with solid tumours.
Time Frame: First treatment cycle, the first 21 days following the start of trial medication.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 9 | 9 | 9 | 9 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Dose Expansion: Number of Patients With Objective Response (OR) - Confirmed Complete Response (CR) and Partial Response (PR)
Description: Dose expansion: Number of patients with objective response (OR) - confirmed complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 as assessed by the Investigator during the entire treatment.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period), up to 818 days.
Population: The Treated Set (TS) included all patients in the dose expansion cohort who received at least 1 dose of BI 754111 or ezabenlimab and had a post baseline measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Dose-Expansion Cohort J: 600 milligram (mg) BI 754111 and 240 mg ezabenlimab given as an intravenous infusion on day 1 of 21-day cycles (q3w) patients with 1st line epidermal growth factor receptor (EGFR) wildtype (WT) and anaplastic lymphoma kinase (ALK) wildtype NSCLC. Patients may have any level of PD-L1 expression, but only a maximum of 10 patients with PD-L1 high expression (=50% PD-L1) were enrolled.
Arm/Group | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Number analyzed (Participants) | 18 | 36 | 37 | 15
Participants | 0 | 3 | 4 | 3

4. Secondary Outcome: Dose Escalation: Number of Patients With Objective Response (OR) - Confirmed Complete Response (CR) and Partial Response (PR)
Description: Dose escalation: Number of patients with objective response (OR) - confirmed complete response (CR) and partial response (PR) according to RECIST Version 1.1 as assessed by the Investigator during the entire treatment.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period), up to 1286 days.
Population: The Treated Set (TS) included all patients in the dose escalation cohort who received at least 1 dose of BI 754111 or ezabenlimab and had a post baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 7 | 9 | 9 | 9 | 8 | 6
Participants | 0 | 0 | 0 | 2 | 0 | 1 | 1

5. Secondary Outcome: Dose Escalation: Number of Patients Experiencing DLTs
Description: Dose escalation: Number of patients experiencing DLTs from start of treatment until end of treatment (in all cycles).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 9 | 9 | 9 | 9 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Dose Expansion: Duration of Response
Description: Duration of response is measured from the time measurements criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: From the date of objective response until first date that recurrent or PD has been documented, up to 100 weeks.
Population: The Treated Set (TS) included all patients in the dose expansion cohort who received at least 1 dose of BI 754111 or ezabenlimab and had a post baseline measurement and had an objective response.
Measure: Median (Standard Deviation); unit: Weeks
Arm/Group | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Number analyzed (Participants) | 0 | 3 | 4 | 3
Weeks |  | 41.14 (31.74) | 45.93 (31.37) | 21.57 (49.22)

7. Secondary Outcome: Dose Expansion: Percentage of Patients With Disease Control
Description: Dose expansion: Percentage of patients with disease control (CR, PR, or stable disease (SD) according to RECIST Version 1.1) as assessed by the Investigator.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Number analyzed (Participants) | 18 | 36 | 37 | 15
Percentage of participants | 44.4 [21.5 to 69.2] | 38.9 [23.1 to 56.5] | 43.2 [27.1 to 60.5] | 86.7 [59.5 to 98.3]

8. Secondary Outcome: Dose Expansion: Progression-free Survival (PFS)
Description: Dose expansion: Progression-free survival (PFS) is defined as time from first drug intake until disease progression or death from any cause, whichever occurs earlier. The date of progression will be based on the Investigator assessment according to RECIST 1.1.
  For patients with 'event' as an outcome for PFS:
  • PFS [days] = date of outcome - date of start of treatment + 1
  For patients with 'censored' as an outcome for PFS:
  • PFS (censored) [days] = date of outcome - date of start of treatment + 1
  Days were converted into months for reporting.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Number analyzed (Participants) | 21 | 40 | 39 | 17
Months | 2.3 [1.4 to 5.7] | 1.4 [1.3 to 2.8] | 1.5 [1.3 to 4.1] | 5.5 [2.7 to 13.7]

9. Secondary Outcome: Dose Expansion: Number of Patients Experiencing DLTs
Description: Dose expansion: Number of patients experiencing DLTs from start of treatment until end of treatment.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
Number analyzed (Participants) | 21 | 40 | 39 | 17
Participants | 1 | 0 | 0 | 0

10. Secondary Outcome: Dose Escalation: AUC0-504: Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: AUC0-504: area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours.
Time Frame: Within 1 hour before and 1, 4, 7, 24, 72, 168, 336 and 504 hours following the start of infusion in the first treatment cycle.
Population: All patients in the TS who provided at least one evaluable observation for at least one Pharmacokinetic (PK) endpoint and no PK relevant protocol deviations. Only patients in the dose escalation cohort with non-missing data were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hours/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 8 | 9 | 9 | 9 | 9 | 6
microgram*hours/milliliter | 12300 (19.3) | 15700 (17.6) | 14300 (16.8) | 15500 (33.0) | 13600 (16.3) | 15600 (24.7) | 14300 (31.0)

11. Secondary Outcome: Dose Escalation: AUC0-504 Steady State: Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: AUC0-504 steady state: area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours at steady state.
Time Frame: Within 1 hour before and 1, 4, 7, 24, 72, 168, 336 and 504 hours following the start of infusion in the fourth treatment cycle.
Population: All patients in the TS who provided at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviations. Only patients in the dose escalation cohort with non-missing data were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hours/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 4 | 3 | 3
microgram*hours/milliliter | NA (na) — Parameter could not be calculated for less than 2 subjects | 23800 (31.1) | NA (na) — Parameter could not be calculated for less than 2 subjects | 27800 (29.1) | 27000 (36.4) | 22400 (41.2) | 35200 (11.2)

12. Secondary Outcome: Dose Escalation: AUC0-504: Area Under the Concentration-time Curve of BI 754111 in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: AUC0-504: area under the concentration-time curve of BI 754111 in plasma over the time interval from 0 to 504 hours.
Time Frame: as for outcome 10
Population: All patients in the TS who provided at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviations. Only patients in the dose escalation cohort with non-missing data who had enough data to calculate the endpoint were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hours/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 9 | 7 | 9 | 9 | 9 | 6
microgram*hours/milliliter | NA (NA) — below the level of detection | NA (NA) — below the level of detection | 3180 (19.9) | 10000 (31.8) | 18500 (19.5) | 30700 (28.1) | 38100 (30.4)

13. Secondary Outcome: Dose Escalation: AUC0-504 Steady State: Area Under the Concentration-time Curve of BI 754111 in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: AUC0-504 steady state: area under the concentration-time curve of BI 754111 in plasma over the time interval from 0 to 504 hours at steady state.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hours/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 4 | 3 | 3
microgram*hours/milliliter | NA (NA) — Parameter could not be calculated for less than 2 subjects. | NA (NA) — below the level of detection | NA (na) — Parameter could not be calculated for less than 2 subjects. | 14300 (35.6) | 25600 (42.7) | 44900 (32.4) | 83500 (3.58)

14. Secondary Outcome: Dose Escalation: Cmax: Maximum Measured Concentration of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: Cmax: maximum measured concentration of ezabenlimab in plasma over the time interval from 0 to 504 hours.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 9 | 9 | 9 | 9 | 9 | 6
microgram/milliliter | 67.2 (29.5) | 76.8 (19.7) | 69.9 (24.0) | 85.5 (56.9) | 71.2 (17.6) | 76.2 (20.6) | 75.9 (12.2)

15. Secondary Outcome: Dose Escalation: Cmax Steady State: Maximum Measured Concentration of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: Cmax steady state: maximum measured concentration of ezabenlimab in plasma over the time interval from 0 to 504 hours at steady state.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 1 | 2 | 6 | 6 | 5 | 3 | 5
microgram/milliliter | NA (na) — Parameter could not be calculated for less than 2 subjects | 90.6 (26.6) | 96.3 (28.2) | 108 (31.3) | 110 (20.5) | 94.2 (44.9) | 102 (26.9)

16. Secondary Outcome: Dose Escalation: Cmax: Maximum Measured Concentration of BI 754111 in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: Cmax: maximum measured concentration of BI 754111 in plasma over the time interval from 0 to 504 hours.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 4 | 9 | 9 | 9 | 9 | 9 | 6
microgram/milliliter | 1.05 (23.5) | 6.23 (15.7) | 23.5 (20.7) | 67.9 (53.9) | 114 (23.8) | 177 (26.6) | 232 (19.8)

17. Secondary Outcome: Dose Escalation: Cmax Steady State: Maximum Measured Concentration of BI 754111 in Plasma Over the Time Interval From 0 to 504 Hours
Description: Dose escalation: Cmax steady state: maximum measured concentration of BI 754111 in plasma over the time interval from 0 to 504 hours at steady state.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab
Number analyzed (Participants) | 1 | 2 | 6 | 6 | 5 | 3 | 5
microgram/milliliter | NA (na) — Parameter could not be calculated for less than 2 subjects | 3.98 (0.711) | 26.5 (18.0) | 72.2 (31.6) | 142 (24.2) | 220 (32.5) | 294 (23.1)

ADVERSE EVENTS:
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period), up to 1286 days.
Description: The Treated Set (TS) included all patients who received at least 1 dose of BI 754111 or ezabenlimab.
Arm/Group | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab | Dose-Expansion Cohort G | Dose-Expansion Cohort H | Dose-Expansion Cohort I | Dose-Expansion Cohort J
All-Cause Mortality (participants affected / at risk) | 0/4 | 3/9 | 2/9 | 1/9 | 2/9 | 3/9 | 0/6 | 16/21 | 27/40 | 25/39 | 11/17
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/9 | 1/9 | 1/9 | 4/9 | 2/9 | 2/6 | 8/21 | 16/40 | 21/39 | 8/17
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 9/9 | 8/9 | 9/9 | 9/9 | 6/6 | 18/21 | 39/40 | 36/39 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab (N=4) | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab (N=6) | Dose-Expansion Cohort G (N=21) | Dose-Expansion Cohort H (N=40) | Dose-Expansion Cohort I (N=39) | Dose-Expansion Cohort J (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort: BI 754111 4 mg + 240 mg Ezabenlimab (N=4) | Dose Escalation Cohort: BI 754111 20 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 80 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 200 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 400 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 600 mg + 240 mg Ezabenlimab (N=9) | Dose Escalation Cohort: BI 754111 800 mg + 240 mg Ezabenlimab (N=6) | Dose-Expansion Cohort G (N=21) | Dose-Expansion Cohort H (N=40) | Dose-Expansion Cohort I (N=39) | Dose-Expansion Cohort J (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 3 | 4 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 5 | 3 | 3
Thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 7 | 4 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2 | 4 | 1 | 3 | 12 | 9 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 1 | 5 | 0 | 4 | 7 | 7 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2 | 3 | 0 | 3 | 8 | 8 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 2 | 2 | 4 | 3 | 3 | 6 | 16 | 17 | 4
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 5 | 9 | 5 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 8 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 3 | 4 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 2 | 3 | 1 | 1 | 3 | 8 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 2 | 3 | 3 | 0 | 4 | 7 | 11 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 3 | 3 | 8 | 5
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 9 | 7 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 7 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 7 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 4 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 3 | 4 | 6 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device malfunction (Product issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 8 | 4 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0 | 2 | 1 | 4 | 5 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 3 | 2 | 1 | 5 | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03156114/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03156114/SAP_001.pdf